CLINICAL TRIAL: NCT05573295
Title: Evaluation of Dental Age of Children With Cleft Lip and Palate Using Willems Method, Cameriere European Formula, and London Atlas
Brief Title: Dental Age Estimation by Different Methods in Patients With Cleft Lip and Palate
Status: Recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yelda Kasımoğlu, Principal investigator, Istanbul University
Other Study IDs: 2021/68
Record Dates: First submitted 2022-10-07; First posted 2022-10-10 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-03

CONDITIONS: Dental Age Estimation; Cleft Lip and Palate
Keywords: children; dental age estimation; Cleft Lip and Palate; chronological age; London Atlas; Cameriere European Formula; Willems method
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with CLP
  Interventions: Other: Diagnostic Test: Willems method; Other: Diagnostic Test: Cameriere method; Other: Diagnostic Test: London Atlas method
- Healthy controls with gender-age match
  Interventions: Other: Diagnostic Test: Willems method; Other: Diagnostic Test: Cameriere method; Other: Diagnostic Test: London Atlas method

INTERVENTIONS:
Other: Diagnostic Test: Willems method — Willems method measures the developmental stages of the seven left permanent mandibular teeth and is frequently used for dental age estimation. The score of each stage is allocated, and the sum of the scores provides an evaluation of the subject's dental maturity.
Other: Diagnostic Test: Cameriere method — Cameriere et al. designed a quantitative approach through a formula based on sex and the ratio between length and apex opening measurements of each lower left tooth.
Other: Diagnostic Test: London Atlas method — The London Atlas requires the user to assess the tooth development and eruption and then match it to one of the 31 pictures of age categories.

SUMMARY:
The aim of this study is to investigate whether there is a significant difference in dental age between children with CLP and healthy controls using the Willems method, Cameriere European formula and London Atlas. It is aimed to create a new formula if there is a significant difference in dental age between children with CLP and healthy controls.

DETAILED DESCRIPTION:
Dental age is widely evaluated by pedodontists, forensic dentists and orthodontists. While a delay in tooth development may be associated with growth retardation and learning difficulties, dental age determination can also be used for forensic age determination for children whose birth information is uncertain. A clear assessment of maturation in children with continued growth is important in establishing a dental treatment plan.

There are two basic approaches to dental age determination in children:

evaluation of eruption of teeth in the oral cavity, evaluation of the development and mineralization of crowns and roots on dental radiographs.

In many methods, the developmental stages of different numbers of permanent teeth are used.

The most commonly used method for determining dental age in children; is the Demirjian method that evaluates the development of seven left permanent mandibular teeth in eight stages (from A to H). Willems et al. In 2001, they modified the Demirjian method by conducting a study on the fact that it showed higher age determination in the Belgian Caucasian population. The adapted method was named the Willems method. It is stated that one of the advantages of this method is that it is a relatively simple system for determining tooth age.

One of the most widely used methods of dental age determination recently is the European formula of Cameriere et al., which is calculated based on open apex. It has been reported that this method has been tested on different population groups, and the results are accurate and reliable.

An atlas method was proposed by a group of London researchers in 2010. The Atlas shows all the teeth array images of certain age groups as a schematic series. Age determination is made by deciding which reference image matches the individual's panoramic radiography image more.

ELIGIBILITY:
Inclusion Criteria:

* 5-14 years old
* Healthy children
* Children with CLP
* Patients without missing left mandibular permanent teeth on panoramic radiography

Exclusion Criteria:

* Children younger than 5 years old and older than 14 years (children that cannot be assessed by the Willems and Cameriere method)
* Poor quality panoramic radiography
* Patients who have received orthodontic treatment
* Patients who received restorative or endodontic treatment

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study was conducted on gender-age matched healthy control group of children aged 5-14 years, who applied to Istanbul University Faculty of Dentistry, Department of Pedodontics, had an AI record in their anamnesis, had panoramic radiographs in the archive of the Department of Oral and Maxillofacial Radiology, Istanbul University Faculty of Dentistry.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient of Willems method | day 1
  Dental age of children with Cleft Lip and Palate and healthy controls assessed by the correlation coefficient
Correlation coefficient of London Atlas method. | day 1
  Dental age of children with Cleft Lip and Palate and healthy controls assessed by the correlation coefficient.
Correlation coefficient of Cameriere European formula. | day 1
  Dental age of children with Cleft Lip and Palate and healthy controls assessed by the correlation coefficient.

SECONDARY OUTCOMES:
Dental age estimation in children with Cleft Lip and Palate | day 1
  Dental age estimation in Turkish children

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No